CLINICAL TRIAL: NCT01255358
Title: Evaluations of Effects of Intra-Erythrocyte Dexamethasone Sodium Phosphate on Neurological Symptoms in Ataxia Teleangiectasia Patients
Brief Title: Intra-Erythrocyte Dexamethasone Sodium Phosphate in Ataxia Teleangiectasia Patients
Acronym: IEDAT-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quince Therapeutics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEDAT-01; 2010-022315-19 (EudraCT Number)
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Nervous System Disorder; Genetic Syndrome
Keywords: Ataxia Teleangiectasia; AT; ERY-DEX; Dexamethasone; Dexamethasone sodium phosphate
MeSH Terms: conditions — Nervous System Diseases; Genetic Diseases, Inborn | interventions — Dexamethasone; dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ERY-DEX (Experimental): Patients treated with monthly treatment of ERY-DEX (dexamethasone sodium phosphate encapsulated in autologous erythrocytes)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone sodium phosphate (2 vials, 250 mg/10 ml each) to be administered via encapsulation into autologous erythrocytes (ERY-DEX system). Final amount administered to the patient: about 10-15 mg of dexamethasone sodium phosphate, encapsulated into autologous blood (2 vials of 250 mg each of dexamethasone sodium phosphate will be used in the ex vivo process together with 50 ml of blood previously taken from the same patient).
  The treatment has to be repeated at intervals of 30 days (±10 days)
  Other Names: Dexamethasone sodium phosphate; Dex 21P

SUMMARY:
The study has the aim to evaluate the improvement in CNS symptoms measured by International Co-operative Ataxia Rating Scale (ICARS) in patients with ataxia teleangectasia (AT), during a period of treatment with ERY-DEX (dexamethasone sodium phosphate ex vivo encapsulated into human autologous erythrocytes).

DETAILED DESCRIPTION:
This is a multi-centre, single arm, open label, 6 months, phase II study to evaluate the effect of ERY-DEX in improving Central Nervous System (CNS) symptoms in patients with Ataxia Teleangectasia (AT). The study consists of a screening period (max duration of 30 days) and a treatment period (duration 6 months).

ELIGIBILITY:
Inclusion Criteria:

* neurological signs of AT
* patients in autonomous gait or helped by a support
* proven molecular diagnosis of AT
* Males and females aged > 3 years
* Body weight >15 kg
* Plasma levels of Lymphocytes CD4+/mm3 > 500 (for patients aged 3-6 years) or > 200 (older than 6 years)
* written IC to participate.

Exclusion Criteria:

* Current or previous neoplastic disease
* History of severe impairment of the immunological system
* Chronic conditions representing a contraindication to the use of steroid drugs
* Non compliance with the study request
* Any previous steroid assumption within 30 days before starting ERY-DEX
* Have any other significant disease that in the Investigator's opinion would exclude the patient from the trial
* Females of childbearing potential who were pregnant, breast-feeding or were not using adequate contraceptive methods

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Chessa, MD, Principal Investigator — A.O. Sant'Andrea Rome Italy
Locations (2):
- Italy (2):
  - Spedali Civili, Brescia
  - University La Sapienza, Rome

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was carried out in 2 Italian Hospitals. Recruitment started on February 2011 and LPLV was performed on August 2011.
Pre-assignment Details: Patients had 30 days of wash-out from steroid assumption before starting the treatment. 26 patients were screened, 4 of them resulted screening failure, due to lymphocytes value below the limit (3) and concomitant disease (1).
Groups:
- EryDex: Patients treated with monthly treatment of EryDex (dexamethasone sodium phosphate encapsulated in autologous erythrocytes).
Period: Overall Study
Arm/Group | EryDex
Started | 22
Completed | 18
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: The study enrolled 22 patients, 11 male and 11 female with a mean age of 11.2. All the enrolled patients received a monthly treatment of EryDex for 6 consecutive months.
Arm/Group | ERY-DEX
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Region of Enrollment [Number; unit: participants]
  Italy | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Neurological Symptoms Assessed by Using International Cooperative Ataxia Rating Scale (ICARS) Score - ITT Population
Description: ICARS ia a 100-point semiquantitative scale, which goes from 0 to 100, offering a compartimentalised quantification of 4 subscores: Posture and Gait Disturbances (maximum score = 34), Kinetic Functions (maximum score = 52), Speech Disorders (maximum score = 8), and Oculomotor Disorders (maximum score = 6) for a possible total score of 100 points. The minimum score is 0 (normal), while the maximum score is 100 and corresponds to the worst status of the patient. This means that for each subscale, higher scores indicate higher levels of impairment.
Time Frame: At visits 2 (day 30), 4 (day 90) and 7 (final visit, day 180)
Population: Intent to treat population (ITT) patients receiving at least one treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ERY-DEX: Patients treated with monthly treatment of ERY-DEX (dexamethasone sodium phosphate encapsulated in autologous erythrocytes)
  Dexamethasone sodium phosphate (2 vials, 250 mg/10 ml each) to be administered via encapsulation into autologous erythrocytes (ERY-DEX system). Final amount administered to the patient: about 10-15 mg of dexamethasone sodium phosphate, encapsulated into autologous blood (2 vials of 250 mg each of dexamethasone sodium phosphate will be used in the ex vivo process together with 50 ml of blood previously taken from the same patient).
  The treatment has to be repeated at intervals of 30 days (±10 days)
Arm/Group | ERY-DEX
Number analyzed (Participants) | 22
units on a scale
  V2 | -2.2 (5.6)
  V4 | -3.4 (7.3)
  V7 | -4.0 (7.5)
Statistical Analysis 1: Comparison: ERY-DEX; The primary analysis on ICARS Total score has been conducted on the ITT Population employing carry-forward and carry-backward procedures for missing data imputation, in order to evaluate all enrolled patients; Test type: Other — Changes from baseline (V1) at V2, V4 and V7 were analyzed with a RMANOVA design with age and ICARS at baseline as covariates. A Wilcoxon non-parametric test between visits was performed when the overall analysis was significant in order to help determine timing of effects; p = 0.02, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-7.1 to -0.9], Standard Deviation 7.5

2. Primary Outcome: Mean Change From Baseline in Neurological Symptoms Assessed by Using International Cooperative Ataxia Rating Scale (ICARS) Score - PP Population
Description: as for outcome 1
Time Frame: At visits 2 (day 30), 4 (day 90) and 7 (final visit, day 180)
Population: The PP Population includes 18 patients who have been treated according to protocol and fulfill the following criteria:
  * compliance with all entry criteria
  * absence of major protocol violations
  * adequate compliance with trial medication (at most one missed or out-of-window infusion of the study preparation).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ERY-DEX
Number analyzed (Participants) | 18
units on a scale
  V2 | -2.4 (4.9)
  V4 | -3.9 (7.1)
  V7 | -5.2 (7.0)
Statistical Analysis 1: Comparison: ERY-DEX; Overall analysis on the PP Population; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0031, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -5.2, 95% CI 2-sided [-8.4 to -2], Standard Deviation 7.0

3. Secondary Outcome: Change From V4 to V7 in Investigator Global Assessment (IGA) - ITT Population
Description: An evaluation of the global health status of the patients by the IGA was performed. IGA consisted of an evaluation of neurological signs and symptoms as neuromotor disorders, posture and deambulation, disturbances of the oro-pharyngeal apparatus, presence of peripheral neuropathy, neurodevelopmental disturbances, intellectual level, and behavior disturbances based only on a subjective judgment of the Investigator on a single scale: a 5-point qualitative scale as:
  * very much improved (1),
  * slightly improved (2),
  * no change (3),
  * slightly worsened (4),
  * very much worsened (5) was used to assess changes from V4 to V7. The higher the score, the worse the outcome.
Time Frame: At visit 7 (final visit, day 180)
Population: The ITT Population includes all 22 patients enrolled into the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ERY-DEX: Patients treated with monthly treatment of ERY-DEX (dexamethasone sodium phosphate encapsulated in autologous erythrocytes).
  Dexamethasone sodium phosphate (2 vials, 250 mg/10 ml each) to be administered via encapsulation into autologous erythrocytes (ERY-DEX system). Final amount administered to the patient: about 10-15 mg of dexamethasone sodium phosphate, encapsulated into autologous blood (2 vials of 250 mg each of dexamethasone sodium phosphate will be used in the ex vivo process together with 50 ml of blood previously taken from the same patient). "
  The treatment has to be repeated at intervals of 30 days (±10 days)
Arm/Group | ERY-DEX
Number analyzed (Participants) | 22
units on a scale | 0.2 (0.6)

4. Secondary Outcome: Change From V4 to V7 in Investigator Global Assessment (IGA) - PP Population
Description: as for outcome 3
Time Frame: At visit 7 (final visit, day 180)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ERY-DEX: Patients treated with monthly treatment of ERY-DEX (dexamethasone sodium phosphate encapsulated in autologous erythrocytes).
  Dexamethasone sodium phosphate (2 vials, 250 mg/10 ml each) to be administered via encapsulation into autologous erythrocytes (ERY-DEX system). Final amount administered to the patient: about 10-15 mg of dexamethasone sodium phosphate, encapsulated into autologous blood (2 vials of 250 mg each of dexamethasone sodium phosphate will be used in the ex vivo process together with 50 ml of blood previously taken from the same patient).
  The treatment has to be repeated at intervals of 30 days (±10 days)
Arm/Group | ERY-DEX
Number analyzed (Participants) | 18
units on a scale | 0.2 (0.6)

5. Secondary Outcome: Mean Change From V4 to V7 in Ocular Motility - ITT Population
Description: An evaluation of ocular motility measured by an ad hoc form was performed at V4 and V7.
  At V4 and V7, ocular motility was assessed through a 5-point qualitative scale: very much improved (1), slightly improved (2), no change (3), slightly worsened (4), very much worsened (5).
Time Frame: At visit 7 (final visit, day 180)
Population: The ITT Population includes all 22 patients enrolled into the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ERY-DEX
Number analyzed (Participants) | 22
units on a scale | -0.3 (0.5)

6. Secondary Outcome: Mean Change From V4 to V7 in Ocular Motility - PP Population
Description: as for outcome 5
Time Frame: At visit 7 (final visit, day 180)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ERY-DEX
Number analyzed (Participants) | 18
units on a scale | -0.3 (0.5)

7. Secondary Outcome: Change From Baseline for Vineland Adaptive Behaviour Scale (VABS) Total Score - ITT Population
Description: VABS aggregate scale is used.
  VABS is divided into 4 adaptive domains and 11 subdomains:
  1. Communication: Receptive, Expressive, Written;
  2. Daily Living Skills: Personal, Domestic, Community;
  3. Socialisation: Interpersonal Relationships, Play & Leisure Time, Coping Skills;
  4. Motor Skills: Gross, Fine.
  For each *question* in each of the 11 subdomains, score ranges from 0 to 4 (the higher the value the better the outcome):
  * 0 = the subject never performs the behaviour without help or reminders;
  * 1 = rarely performs (as above);
  * 2 = sometimes performs (as above);
  * 3 = often performs (as above);
  * 4 = almost always performs (as above); The total subdomain score is the sum of each *question* scores and the total domain score is the sum of each subdomains' scores.
  Domains min-max interval scores:
  0-74 Communication, 0-74 Daily Living Skills, 0-62 Socialization, 0-111 Motor Skills, Sum-of-domains score 0-321(the higher the score, the better the outcome)
Time Frame: At visits 4 (90 days) and 7 (180 days, final visit)
Population: The ITT Population includes all 22 patients enrolled into the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ERY-DEX: Patients treated with monthly treatment of ERY-DEX (dexamethasone sodium phosphate encapsulated in autologous erythrocytes)
  Dexamethasone sodium phosphate (2 vials, 250 mg/10 ml each) to be administered via encapsulation into autologous erythrocytes (ERY-DEX system). Final amount administered to the patient: about 10-15 mg of dexamethasone sodium phosphate, encapsulated into autologous blood (2 vials of 250 mg each of dexamethasone sodium phosphate will be used in the ex vivo process together with 50 ml of blood previously taken from the same patient). "
  The treatment has to be repeated at intervals of 30 days (±10 days)
Arm/Group | ERY-DEX
Number analyzed (Participants) | 22
units on a scale
  V4 | 1.0 (0.9)
  V7 | 1.3 (1.3)
Statistical Analysis 1: Comparison: ERY-DEX; VABS total score at V7; Test type: Other — VABS Total score and subscales have been analyzed with a RMANOVA design, using age as covariate (dichotomized as Low- or High-, using median age as threshold); p < 0.0001, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.3, 95% CI 2-sided [0.8 to 1.8], Standard Deviation 1.2

8. Secondary Outcome: Change From Baseline for Vineland Adaptive Behaviour Scale (VABS) Total Score - PP Population
Description: as for outcome 7
Time Frame: At visits 4 (90 days) and 7 (180 days, final visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ERY-DEX
Number analyzed (Participants) | 18
units on a scale
  V4 | 1.1 (0.9)
  V7 | 1.5 (1.1)
Statistical Analysis 1: Comparison: ERY-DEX; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 1.5, 95% CI 2-sided [1 to 2], Standard Deviation 1.1

9. Secondary Outcome: Count of Participants on ERY-DEX Showing Treatment Emergent Adverse Events (TEAEs) Including Serious Adverse Events (SAEs)
Description: The effect of ERY-DEX on treatment emergent adverse events was expressed as the number of patients showing at least one TEAE or 1 serious AE
Time Frame: Throughout the study, until the end of 6 months of treatment (day 180)
Population: The SP includes the 22 patients who have received at least one dose of planned trial treatment.
Measure: Count of Participants; unit: Participants
Groups:
- ERY-DEX: Patients treated with monthly treatment of EryDex (dexamethasone sodium phosphate encapsulated in autologous erythrocytes)
  dexamethasone sodium phosphate (2 vials, 250 mg/10 ml each) to be administered via encapsulation into autologous erythrocytes (ERY-DEX system). Final amount administered to the patient: about 10-15 mg of dexamethasone sodium phosphate, encapsulated into autologous blood (2 vials of 250 mg each of dexamethasone sodium phosphate will be used in the ex vivo process together with 50 ml of blood previously taken from the same patient).
  The treatment has to be repeated at intervals of 30 days (±10 days)
Arm/Group | ERY-DEX
Number analyzed (Participants) | 22
Participants
  Participants with at least 1 TEAE | 15
  Participants with at least 1 serious AE | 2

ADVERSE EVENTS:
Time Frame: The adverse events were monitored and collected during the 6 month study period
Description: Please note that non serious Adverse Events were monitored/assessed without regard to the specific Adverse Event Term but only by SOC.
Arm/Group | Ery-Dex
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 15/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ery-Dex (N=22)
Bronchopneumonia (Infections and infestations) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ery-Dex (N=22)
General disorders (General disorders) | 3 (3)
immune disorders (Immune system disorders) | 2 (2)
infections and infestations (Infections and infestations) | 15 (17)
respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less